CLINICAL TRIAL: NCT01060761
Title: Involvement of Patients and Relatives in the Course of Cancer Disease With a Particular View to Rehabilitation and the Life With Cancer
Brief Title: Involvement of Patients and Relatives in the Course of Cancer Disease
Acronym: KRIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Helle Ploug Hansen, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HMS-SDU- 2009-1
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2012-06

CONDITIONS: Rehabilitation; Cancer; Relatives
Keywords: cancer; Rehabilitation program (patient and a relative together); counselling; retreat weekend
MeSH Terms: conditions — Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation program (Active Comparator): Counselling (supportive conversation with patient and their relatives together) Retreat Weekend (patient and their relatives together)
  Interventions: Behavioral: Rehabilitation program
- Ususal treatment and support (No Intervention): Usual support and treatment at the hospital, no retreat Weekend.

INTERVENTIONS:
Behavioral: Rehabilitation program — Patient and their relative receive three supportive, structured conversation with a trained nurse.
  Patient and their relative receive 4 days Retreat Weekend with supportive talk and activities
  Other Names: KRIPP project
  Arms: Rehabilitation program

SUMMARY:
The objective is to investigate a rehabilitation program (supportive conversations and a rehabilitation course for cancer patients and their relatives together).

The study evaluate the effect of the program compared to no intervention (usual care)

DETAILED DESCRIPTION:
The study aim to evaluate the effect and the benefit of the program.

First the patients psychosocial well-being is assessed in a survey (EORTC, POMS, WHO-5 well-being index) Then their relatives psychosocial well-being is assessed in a survey (Ad hoc questions, POMS and WHO-5 well-being index)

The effect is also assessed in qualitative interviews with patients and their relatives.

The rehabilitation course is investigated in qualitative observations and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Both the patient and their relative must agree to participate together
* Patient admitted to the Hospital
* Patient admitted with a lung cancer diagnosis or
* Patient admitted with a gynecological cancer diagnosis

Exclusion Criteria:

* The cancer diagnosis was not verified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Quality of life, | two months and one year

CONTACTS AND LOCATIONS:
Overall Officials: Helle P Hansen, Professor, Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark